CLINICAL TRIAL: NCT06033365
Title: Beginning Early and Assertive Treatment for Methamphetamine Use Disorder (BEATMeth): A Comprehensive Systems-level Secondary Prevention Strategy to Prevent Stimulant Related Overdoses
Brief Title: Beginning Early and Assertive Treatment for Methamphetamine Use Disorder
Acronym: BEATMeth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Denver Health and Hospital Authority (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 22-0968; R01CE003363 (NIH)
Record Dates: First submitted 2023-04-25; First posted 2023-09-13 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-11

CONDITIONS: Methamphetamine Use Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Dedicated care navigator to address social support needs
  Interventions: Behavioral: care navigation
- Usual care (No Intervention): Standard of care.

INTERVENTIONS:
Behavioral: care navigation — Dedicated care navigation throughout study enrollment and follow-up period. Care navigation consists of addressing social support needs (e.g. transportation, communication, housing).
  Arms: Intervention

SUMMARY:
The overall goal of the study is to evaluate the effectiveness of a secondary prevention strategy implemented at a systems-level to prevent stimulant related overdoses.

DETAILED DESCRIPTION:
To date, a public health systems approach to enhance linkage and engagement in care for stimulant use disorders is lacking. This shortcoming arises in part from the lack of effective treatments for stimulant use disorders (StUD), the specific pathology of methamphetamine use, and gaps in epidemiologic knowledge related to methamphetamine use disorder. Unlike opioid use disorders, for which medications relieve dysphoric symptoms of acute withdrawal and prevent relapse, patients with StUD present to care with methamphetamine-induced psychosis and may be combative, agitated, and poorly insightful to their need for treatment. In response to community demands, our team at Denver Health recently established a pilot program, Beginning Early and Assertive Treatment for Methamphetamine Use Disorder (BEAT Meth), to protocolize the assessment and treatment of patients with methamphetamine-induced psychosis.The current research project aims to develop and conduct process and outcomes evaluations of a linkage intervention aimed at increasing continuation and engagement in treatment for stimulant use disorder.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and older
* identified in the Denver Health healthcare system who have had a methamphetamine-related encounter at Denver Health

Exclusion Criteria:

* unable to complete the interview in English
* intoxicated or impaired and unable to consent to participate in the project and/or respond to the interview
* currently under residential involuntary psychiatric or substance treatment order (i.e., mental health hold, emergency commitment, or short-term certification)
* received any type of substance use treatment at DHHA in the last 90 days
* planning to enter substance treatment
* unable to complete the research visits in the next 90 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 192 (Actual)
Dates: Start 2023-04-11 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-09-29 (Actual)

PRIMARY OUTCOMES:
Number of participants who entered treatment for methamphetamine use disorder | within 30 of study enrollment
  Treatment entry as defined as attendance at an outpatient addiction treatment appointment within 30 days of BEAT Meth discharge

SECONDARY OUTCOMES:
Number of participants retained in treatment at 30 days | 30 days
  Retention in treatment at 30 days
Number of participants who overdosed | through study completion, an average of 1 year
  non-fatal overdose as self-reported and fatal overdose from medical examiner
Number of participants retained in treatment at 90 days | 90 days
  Retention in treatment at 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Alia A Al-Tayyib, PhD, Principal Investigator — Denver Health
Locations (1):
- Denver Health, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2023-04-06): https://cdn.clinicaltrials.gov/large-docs/65/NCT06033365/ICF_000.pdf